CLINICAL TRIAL: NCT02114372
Title: Cognitive Health in Ageing Register: Investigational, Observational and Trial Studies in Dementia Research (CHARIOT): Prospective Readiness Cohort Study (PRO)
Brief Title: Cognitive Health in Ageing Register: Investigational, Observational and Trial Studies in Dementia Research: Prospective Readiness Cohort Study
Acronym: CHARIOT:PRO
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR104383; REGISTRYALZ0001; RRA-11823 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-04-11; First posted 2014-04-15 (Estimated); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer's Disease; Plaque, Amyloid
Keywords: Alzheimer's disease; Asymptomatic at risk for Alzheimer's disease; Retinal diagnosis for Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva, and urine specimens will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CogState Brief Battery: Enrolled participants will be randomized in a balanced manner to CogState brief battery in both the Main Study and the SubStudy. CogState consists of four tasks that respectively measure the functions of attention, processing speed, visual learning, and working memory. The CogState Brief Battery is an approximately 15 minute computerized battery with demonstrated reliability, validity, and short term stability, that was developed expressly for maximal sensitivity to detect change. CogState can be administered via the internet or on a stand-alone computer and is available in over 50 languages.
- Cognitive Drug Research Assessment System (CDR-AS): Enrolled participants will be randomized in a balanced manner to CDR-AS in both the Main Study and the SubStudy. CDR-AS is fully automated system that targets the core aspects of cognitive function crucial for everyday behavior which are vulnerable to numerous insults including aging, fatigue, disease, pathology, trauma, diet, and pharmaceuticals. CDR-AS is an approximately 20-minute computerized battery designed to reliably measure changes in cognitive function in clinical trial situations.
- Delis Kaplan Executive Function System (DKEFS): Enrolled participants will be randomized in a balanced manner to DKEFS in the Main Study and at one site of the SubStudy. The DKEFS is a paper and pencil measure of verbal and nonverbal executive functions that has been normed and validated for children and adults from 8-89 years of age. The measure consists of nine subtests. For the purposes of this study, the Trail Making Test (TMT) and Verbal Fluency subtests will be used.
- COGNITO: Enrolled participants will be randomized in a balanced manner to COGNITO at the other site of the SubStudy. COGNITO is an approximately 45 to 60 minute computerized neuropsychometric examination based on well-known cognitive tests designed for both cognition research and clinical assessment. COGNITO assesses reaction time, primary and working memory, visuospatial and verbal secondary memory, implicit learning, language skills, functional and semantic categorization of visual data, focused and divided attention, and crystallized intelligence. Responses are made via a tactile screen which permits the recording of response latency (deducting reaction time provides an estimation of information processing time).

SUMMARY:
The purpose of this study is to prospectively investigate the longitudinal change of the components of the Preclinical Alzheimer Cognitive Composite (PACC) and the components (index scores) of the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) in asymptomatic at risk for Alzheimer's disease (ARAD) individuals.

DETAILED DESCRIPTION:
This is a prospective, non-interventional study that will enroll participants without dementia who are considered at high, medium, and low risk for developing AD from a community based register (referred to as the CHARIOT registry) in the United Kingdom. Participants will undergo a series of neuropsychological evaluations to characterize the patterns of cognitive change and their inter-relationship in the earliest stages of cognitive impairment. In addition, how such changes relate to the clinical presentation of cognitive impairment of the Alzheimer's type may be evaluated over time. The SubStudy will investigate the longitudinal change of components of the PACC and RBANS in ARAD individuals who have demonstrable amyloid in the brain by either PET or CSF compared with individuals not classified as ARAD. SubStudy participants will be followed every 6 months throughout the SubStudy and will alternate between completing the alternative forms of the PACC and RBANS for a period of up to 4.5 years (54 months). Blood, urine, and saliva samples will be collected from participants during the study for biomarker analyses to assess risk factors for dementia, Alzheimer's disease or confounding factors of dementia risk. Adverse events experienced by the participants during their participation in the study will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Completed Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) and Preclinical Alzheimer Cognitive Composite (PACC) neurocognitive testing at least once during the SubStudy screening visits
* Have a global Clinical Dementia Rating (CDR) score of 0 at screening
* Be fluent in and able to read and write in English; be willing and able to give written informed consent; and have adequate hearing and visual acuity to complete the required psychometric tests
* Have evidence of amyloid pathology by means of low cerebrospinal fluid (CSF) beta amyloid protein (ABeta42) concentrations at screenings (for amyloid positive cohort only) or have no evidence of amyloid pathology by this criterion (for amyloid negative cohort only) and are selected for inclusion in Cognitive Health in Ageing Register: Investigational, Observational, and Trial studies in dementia research: Prospective Readiness cohort study (CHARIOT-PRO) as per the interactive web response decision algorithm
* Be otherwise in satisfactory health and medically stable on the basis of medical history, vital signs, and physical exam. Any abnormalities must not be the cause or be associated with cognitive impairment

Exclusion Criteria:

* Meets clinical criteria for Alzheimer's disease (AD) dementia, Mild Cognitive Impairment (MCI) diagnosis, or has any degenerative brain disorder that is associated with dementia, such as Parkinson's disease
* Participants whose age- and education-adjusted cognitive performance is more than 1.5 standard deviation (SD) below normal on any of the RBANS Index scores at the first RBANS administration
* Any known history of familial autosomal dominant AD or other familial dementing diseases
* History of or current thyroid disease or thyroid dysfunction, which is currently uncontrolled or untreated, or clinically significant abnormal thyroid function tests. Participants treated for thyroid disease may be enrolled following review of their records of thyroid function, laboratory tests at screening, diagnosis and treatment history by the Investigator or designee
* Any contraindications for magnetic resonance imaging (MRI) (example, pacemaker, metal prostheses, implants, claustrophobia, pacemakers etc) unless MRI compatible

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SubStudy includes participants who have completed Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) and Preclinical Alzheimer Cognitive Composite (PACC) neurocognitive testing at least once during the SubStudy screening visits and have a baseline global Clinical Dementia Rating scale (CDR) score of 0.
Sampling Method: Non-Probability Sample
Enrollment: 1136 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Main Study: Change From Baseline Cognition | Up to 4 years
  Cognition will be evaluated at baseline and longitudinally with the Mini-Mental State Examination (MMSE), Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), Neuropsychological Assessment Battery (NAB)-Executive Function module, NAB-Memory module, CogState Brief Battery (CBB), Cognitive Drug Research Assessment System (CDR-AS), and Delis Kaplan Executive Function System (DKEFS), as well as the Clinical Dementia Rating Scale.
SubStudy: Change From Baseline on Preclinical Alzheimer Cognitive Composite (PACC) Component Score | Baseline and Month 42 (Year 3.5)
  The PACC is a retrospectively validated measure that is weighted towards episodic memory, and also includes a timed executive function test and a global cognitive screening test. The PACC includes: 1. Total Recall score from the Free and Cued Selective Reminding Test - Immediate Recall [FCSRT-IR] (0-48 words); 2. Delayed Paragraph Recall total score on single administration of the Logical Memory story from the Wechsler Memory Scale [WMS]-Revised (0-25 story units); 3. Digit Symbol Substitution Test score from the Wechsler Adult Intelligence Scale [WAIS]-Revised (0-135 symbols), and 4. MMSE score (0-30 points). The component scores are transformed using an established normalization method into z-scores. Each of the 4 component change scores is divided by the baseline sample standard deviation of that component. Z-score implies how many standard deviations higher or lower the score is compared with the baseline score.
SubStudy: Change From Baseline in RBANS Index Scores | Baseline and Month 42 (Year 3.5)
  This brief test is for cognitive assessment, detection, and characterization of dementia in the elderly as well as neuropsychological screening for younger patients. The RBANS Index scores include Immediate Memory Index, Visuospatial/Construction Index, Language Index, Attention Index and the Delayed Memory Index. The sum of these 5 Index scores is converted to a Total Scale value via a mapping table. The Total Scale is a norm-based t score based on a distribution with a mean of 100 and standard deviation of 15.

SECONDARY OUTCOMES:
SubStudy: Change From Baseline on the RBANS Total Scale | Baseline and Month 42 (Year 3.5)
  RBANS is a battery developed for cognitive assessment, detection, and characterization of dementia in the elderly as well as neuropsychological screening for younger patients. The RBANS includes 12 subtests that measure 5 indices: the Attention Index is composed of Digit Span and Coding, the Language Index consists of Picture Naming and Semantic Fluency subtests, the Visuospatial/Construction Index is made up of Figure Copy and Line Orientation subtests, the Immediate Memory Index is composed of List Learning and Story Memory subtests, and the Delayed Memory Index consists of List Recall, List Recognition, Story Recall, and Figure Recall subtests. The sum of these 5 Index scores is converted to a Total Scale value via a mapping table. The Total Scale is a norm-based t score based on a distribution with a mean of 100 and standard deviation of 15.
SubStudy: Change From Baseline on the PACC Composite Score | Baseline and Month 42 (Year 3.5)
  The PACC is retrospectively validated measure that is weighted towards episodic memory, timed executive function test and global cognitive screening test. The PACC includes: 1. Total Recall score from FCSRT-IR (0-48 words); 2. Delayed Paragraph Recall total score on single administration of Logical Memory story from the WMS-Revised (0-25 story units); 3. Digit Symbol Substitution Test score from WAIS-Revised (0-135 symbols), and 4. MMSE score (0-30 points). The composite score is determined from its components using an established normalization method. Each of the 4 component change scores is divided by the baseline sample standard deviation of that component, to form standardized z-scores. Z-score implies how many standard deviations higher or lower the score is compared with baseline score. The composite score is sum of z-scores for component scores. Thus, a change of 1 baseline standard deviation on each component would correspond to a 4-point change on the composite.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United Kingdom (2):
  - Edinburgh
  - London

REFERENCES:
- [Derived] Taylor S, Dunn L, Udeh-Momoh C, Abbott K, Giannakopoulou P, Middleton L, Robinson O, Kalsi J, Kafetsouli D, Ford J. Technology readiness among UK-based cognitively unaffected older adults during the COVID-19 pandemic: potential implications for decentralised alzheimer's disease prevention trials. BMC Geriatr. 2025 Jul 30;25(1):563. doi: 10.1186/s12877-025-06158-3. PMID 40739178
- [Derived] Udeh-Momoh CT, Watermeyer T, Price G, de Jager Loots CA, Reglinska-Matveyev N, Ropacki M, Ketter N, Fogle M, Raghavan N, Arrighi M, Brashear R, Di J, Baker S, Giannakopoulou P, Robb C, Bassil D, Cohn M, McLellan-Young H, Crispin J, Lakey K, Lisa C, Chowdary Seemulamoodi Y, Kafetsouli D, Perera D, Car J, Majeed A, Ward H, Ritchie K, Perneczky R, Kivipelto M, Scott D, Bracoud L, Saad Z, Novak G, Ritchie CW, Middleton L. Protocol of the Cognitive Health in Ageing Register: Investigational, Observational and Trial Studies in Dementia Research (CHARIOT): Prospective Readiness cOhort (PRO) SubStudy. BMJ Open. 2021 Jun 24;11(6):e043114. doi: 10.1136/bmjopen-2020-043114. PMID 34168021